CLINICAL TRIAL: NCT06451016
Title: Effects of Vitamin D Supplementation on Muscle Function Among Grave's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frontier Medical and Dental College, Abbotabad (Other)
Responsible Party: Principal Investigator, Dr Saif ur Rehman, Professor, Frontier Medical and Dental College, Abbotabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3389
Record Dates: First submitted 2024-05-29; First posted 2024-06-10 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Graves Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental)
  Interventions: Dietary Supplement: Vitamin D supplements
- Control Group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D supplements — 70 mcg/day (equal to 2800 IU) of cholecalciferol
  Arms: Vitamin D group
Dietary Supplement: Placebo — Matching Placebo
  Arms: Control Group

SUMMARY:
Introduction:

A deficit in vitamin D may be involved in the development and presentation of Graves' disease (GD). Lack of vitamin D and GD are linked to deteriorating quality of life (QoL) and weakening of the muscles. Our goal was to look at the possible advantages of vitamin D supplementation for the improvement of thyroid-related QoL and muscle function in GD patients, as well as the possible drawbacks of anti-thyroid drugs (ATD).

Methodology:

A multicenter randomized controlled experiment with single-blinding was carried out with 48 patients who had been diagnosed with Graves' illness. The participants were split into two groups n=24 patients in each group. In addition to standard ATD, Group A received either 70 μg (2800 IU) of vitamin D daily or a corresponding placebo. Investigator measured muscular function and isometric strength at baseline, three, and nine months.

ELIGIBILITY:
Inclusion Criteria:

* Grave's Disease
* either starting or about to start anti-thyroid medication (ATD)

Exclusion Criteria:

* Chronic granulomatous disease
* hypercalcemia
* poor renal function (eGFR < 45 ml/min)
* the presence of malignant disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | base line and after 3months
  Hand Grip strength was measured using dynamometer

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Frontier Medical and Dental College, Abbottābād, KPK
  - Frontier Dental, Abbottābād, Sindh